CLINICAL TRIAL: NCT01847703
Title: Randomized Trial Comparing Robotic and Abdominal Surgery for High Risk Endometrial Cancer
Brief Title: Robotic Versus Abdominal Surgery for Endometrial Cancer
Acronym: RASHEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Henrik Falconer, MD, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/361-31/1
Record Dates: First submitted 2013-05-02; First posted 2013-05-07 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Endometrial Neoplasms
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Robotic surgery (Experimental): Experimental method, to be compared with standard care
  Interventions: Procedure: Robotic surgery
- Abdominal surgery (Active Comparator): Conventional open surgery (laparotomy)
  Interventions: Procedure: Abdominal surgery

INTERVENTIONS:
Procedure: Robotic surgery — Minimal invasive surgery performed with daVinci robotic system
  Arms: Robotic surgery
Procedure: Abdominal surgery — Current gold standard
  Arms: Abdominal surgery

SUMMARY:
This study is intended to explore differences in oncologic and surgical safety between robotic assisted laparoscopy and conventional abdominal surgery for high risk endometrial cancer.

DETAILED DESCRIPTION:
Hypothesis: Robotic assisted laparoscopy (RAL)is equal in terms of oncologic and surgical safety as conventional abdominal surgery (AS) for high risk endometrial cancer (EC).

Methods: Women with high risk EC (defined as high grade endometrial, clear cell or serous) are randomized to either RAL or AS. Both groups will undergo complete surgical staging (hysterectomy, bilateral salpingoophorectomy, pelvic and paraaortal lymphadenectomy)

Primary endpoint: Number of harvested lymph nodes per station Secondary endpoints: Recurrences up to 3 year after surgery. Lymphatic side-effects, quality of life, cost, surgical morbidity.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age
* High risk endometrial cancer

Exclusion Criteria:

* WHO performance>1
* Severe comorbidity, ASA>3
* Unable to understand information

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-04; Primary Completion 2016-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Number of harvested lymph nodes | 2 years
  Extracted lymphatic tissue from 3 stations (above inferior mesenteric artery, below inferior mesenteric artery, pelvic) is analysed by a pathologist and the number of nodes for each station recorded and compared between the two groups

SECONDARY OUTCOMES:
Recurrence of cancer | 3 years
  Cancer recurrences will be recorded up to 3 years after surgery and categorized according to anatomical site
Lymphatic side-effects | 2 years
  Lymphatic side-effects will be monitored by repeated computed tomography (CT) 3 months and 12 months after surgery. Enrolled women will be asked specific, validated questions at follow-up
Quality of life | 2 years
  All included participants will be asked to fill out a questionnaire (EORTC) to assess quality of life before and 1 year after surgery
Healthcare cost | 2 years
  All costs related to each procedure including complications, re-admissions, rehabilitation, medication, radiology will be compared after 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Falconer, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Salehi S, Avall-Lundqvist E, Legerstam B, Carlson JW, Falconer H. Robot-assisted laparoscopy versus laparotomy for infrarenal paraaortic lymphadenectomy in women with high-risk endometrial cancer: A randomised controlled trial. Eur J Cancer. 2017 Jul;79:81-89. doi: 10.1016/j.ejca.2017.03.038. Epub 2017 Apr 29. PMID 28463759